CLINICAL TRIAL: NCT04552457
Title: Do Liberal Versus Strict Postoperative Restrictions After Mid-urethral Slings Affect Outcomes?
Brief Title: Postoperative Activity Restrictions After Slings
Acronym: PARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0141
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Stress Urinary Incontinence; Patient Satisfaction; Surgery
Keywords: Mid-urethral sling; Postoperative activity; Activity restriction
MeSH Terms: conditions — Urinary Incontinence, Stress; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No activity restrictions (Experimental)
  Interventions: Behavioral: No activity restrictions
- Activity restrictions (Active Comparator)
  Interventions: Behavioral: Activity restrictions

INTERVENTIONS:
Behavioral: No activity restrictions — Patients in the "No activity restrictions" group will be allowed to return to their normal activity immediately.
  Arms: No activity restrictions
Behavioral: Activity restrictions — Patients in the "Activity restrictions" group will not be allowed to perform strenuous exercise or lift anything greater than 10lbs. "Strenuous exercise" will be defined as is any activity that requires so much exertion that one cannot have a conversation comfortably while doing it.
  Arms: Activity restrictions

SUMMARY:
Postoperative restrictions are often based on expert opinion and "common sense". There is a wide variety in the recommended activity limitation amongst pelvic floor surgeons. Many patients undergo urogynecologic procedures to improve their quality of life, and these additional restrictions decrease their quality of life in the short term. Our hypothesis is that unrestricted activity after a mid-urethral sling will not negatively impact a patient's recovery or likelihood of surgical success.

Eligible participants will be randomized to no postoperative instructions or traditional postoperative instructions. Patients will be followed up at 2 weeks, 6 weeks, and 6 months postoperatively. Data will be collected throughout the follow up period, but the primary endpoint is at 6 months. At the 6 month visit, subjects' activity level, leakage symptoms, and postoperative satisfaction will be assessed.

DETAILED DESCRIPTION:
There is a limited body of literature regarding restrictions for gynecologic surgery. Most of these studies have looked at patients with prolapse and incontinence, and many of the postoperative recommendations are intended for both classes of procedures. Most surgeons restrict their patients' activities postoperatively but to varying degrees and for variable amounts of time. One study in 2017 showed no adverse effect on short term outcomes after prolapse repair with liberal postoperative restrictions compared to stricter, traditional restrictions. No studies have been performed to look at postoperative restrictions after mid-urethral slings.

A common reason for limiting activity is due to the unproven concern about increased intra-abdominal pressure on healing and surgical success. At this time, no studies have shown causality. The range of intra-abdominal pressures generated during "unavoidable" activities, such as coughing, standing, and bending, overlaps with the range of pressures generated during activities that are typically restricted. Another study showed the intra-abdominal pressures generated during activities of daily living overlapped with pressures generated by women performing CrossFit exercises.

A 2017 study showed no effect on outcomes with unrestricted activity after pelvic reconstructive surgery. Orthopedic literature suggests better outcomes with early postoperative activity over immobilization. There is a significant body of literature showing potential detrimental effects of sedentary behavior and bed rest.

In 2010, an estimated 28.1 million women had urinary incontinence; however only 260,000 sling surgeries were performed that year. As stress urinary incontinence is primarily thought to result from a loss of support for the urethra, anatomic repair key to its treatment. Many women delay any type of treatment for stress urinary incontinence due to lack of awareness or belief in the myth that stress incontinence is a "normal part of aging". The arbitrary activity restrictions serve as yet another obstacle to treatment, especially for women who work as physical laborers. Since these activity restrictions are rooted in medical dogma and there is no evidence supporting the necessity of postoperative activity restrictions, this is a significant, iatrogenic barrier to care for all women with stress urinary incontinence. Our study could provide objective evidence of the effects of activity on satisfaction and surgical success after mid-urethral slings.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85 years
* Urodynamic-proven stress incontinence or stress leakage on physical exam
* Desires surgical management for stress incontinence with a midurethral sling

Exclusion Criteria:

* Prior midurethral sling or urethropexy
* Prior pelvic reconstruction
* Prior pelvic radiation
* Connective tissue disorder
* Severe physical limitation at baseline
* Currently pregnant or desires future childbearing potential
* Concomitant surgeries (except for anterior colporrhaphy for anterior wall prolapse less than 0 on POPQ or other minor procedures).

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with postoperative course | 6 months
  5-point scale with minimum of 1 and maximum of 5 points, higher scores corresponding to more satisfaction

SECONDARY OUTCOMES:
Surgical success | 6 months
  Presence of persistent or recurrent stress urinary incontinence as defined as positive cough stress test and positive response on Urogenital Distress Inventory short form.

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Great Neck, New York, United States

REFERENCES:
- [Background] Gephart LF, Doersch KM, Reyes M, Kuehl TJ, Danford JM. Intraabdominal pressure in women during CrossFit exercises and the effect of age and parity. Proc (Bayl Univ Med Cent). 2018 Apr 9;31(3):289-293. doi: 10.1080/08998280.2018.1446888. eCollection 2018 Jul. PMID 29904290
- [Background] Mueller MG, Lewicky-Gaupp C, Collins SA, Abernethy MG, Alverdy A, Kenton K. Activity Restriction Recommendations and Outcomes After Reconstructive Pelvic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Apr;129(4):608-614. doi: 10.1097/AOG.0000000000001924. PMID 28277355
- [Background] Weir LF, Nygaard IE, Wilken J, Brandt D, Janz KF. Postoperative activity restrictions: any evidence? Obstet Gynecol. 2006 Feb;107(2 Pt 1):305-9. doi: 10.1097/01.AOG.0000197069.57873.d6. PMID 16449116
- [Background] McCormack R, Bovard J. Early functional rehabilitation or cast immobilisation for the postoperative management of acute Achilles tendon rupture? A systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2015 Oct;49(20):1329-35. doi: 10.1136/bjsports-2015-094935. Epub 2015 Aug 17. PMID 26281836
- [Background] Nygaard IE, Hamad NM, Shaw JM. Activity restrictions after gynecologic surgery: is there evidence? Int Urogynecol J. 2013 May;24(5):719-24. doi: 10.1007/s00192-012-2026-2. Epub 2013 Jan 23. PMID 23340879
- [Background] FitzGerald MP, S. S., Shott S, Brubaker L (2001).
- [Background] Magon N, Kalra B, Malik S, Chauhan M. Stress urinary incontinence: What, when, why, and then what? J Midlife Health. 2011 Jul;2(2):57-64. doi: 10.4103/0976-7800.92525. PMID 22408333
- [Background] Murphy M. Restrictions and limitations after pelvic floor surgery: what's the evidence? Curr Opin Obstet Gynecol. 2017 Oct;29(5):349-353. doi: 10.1097/GCO.0000000000000393. PMID 28719393
- [Derived] Lai E, McDonald K, Chopra V, Robinson L, Alvarez A, O'Shaughnessy D, Pillalamarri N, Polland A, Shalom D, Winkler H. Postoperative Activity Restrictions After Slings: A Randomized Controlled Trial. Urogynecology (Phila). 2025 Jun 1;31(6):619-626. doi: 10.1097/SPV.0000000000001515. Epub 2024 May 6. PMID 38710013